CLINICAL TRIAL: NCT06951581
Title: A Randomized, Placebo-controlled Trial Investigating the Effect of Short-chain Fatty Acid (SCFA) Supplementation on Serum and Urinary Metabolome in Kidney Transplant Recipients (METAKID Study)
Brief Title: Impact of SCFA Supplementation on Metabolic Profiles in Serum and Urine of Kidney Transplant Recipients.
Acronym: METAKID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Martin (Other)
Collaborators: Comenius University (Other)
Responsible Party: Principal Investigator, Matej Vnucak, deputy head of Transplant-nephrology Department, University Hospital, Martin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TNO_UNM_SCFA1
Record Dates: First submitted 2025-04-08; First posted 2025-04-30 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Effects; Immunosuppressive Agents; Adverse Events; Imunological Effects; Inflamatory Markers; Metabolomic Effects; Renal Function
Keywords: short chain fatty acids; urine and serum metabolomics; kidney transplant recipients
MeSH Terms: interventions — Fatty Acids, Volatile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCFA Group (Active Comparator): Participants will receive an oral formulation of short-chain fatty acids (SCFA) in dose 200 mg daily for 12 weeks
  Interventions: Dietary Supplement: Short Chain Fatty Acid
- Placebo Group (Placebo Comparator): Participants will receive a placebo orally (sacharosis in dose 200 mg), matching the SCFA formulation in appearance and administration schedule, for 12 weeks.
  Interventions: Dietary Supplement: Placebo Capsule(s)

INTERVENTIONS:
Dietary Supplement: Short Chain Fatty Acid — Participants in this arm will receive an oral formulation of short-chain fatty acids (SCFAs) daily for 12 weeks. SCFAs are administered as a dietary supplement to investigate their potential impact on the systemic and urinary metabolome in kidney transplant recipients.
  Arms: SCFA Group
Dietary Supplement: Placebo Capsule(s) — Oral capsules with sacharosa (200 mg) matching SCFA appearance, administered once a day.
  Arms: Placebo Group

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial evaluating the impact of short-chain fatty acid (SCFA) supplementation on the serum and urinary metabolome in stable kidney transplant recipients. A total of eligible patients will be randomized 1:1 to receive either SCFA or placebo for a period of 12 weeks. Metabolomic profiling of serum and urine will be performed at three time points: at baseline, after 12 weeks of intervention, and after a 12-week washout period without supplementation. The primary objective of the study is to investigate whether SCFA supplementation leads to measurable changes in systemic and renal metabolomic profiles. Secondary outcomes include assessment of tolerability, safety, and potential immunometabolic correlations and also impact on the serum level of immunossupresants (tacrolimus). This study aims to explore the potential of microbiota-targeted therapies in modulating post-transplant metabolic homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

Stable kidney transplant recipients (≥ 6 months post-transplantation)

Stable graft function defined as eGFR ≥ 30 mL/min/1.73 m² with no significant change (>15%) in the last 3 months

No episodes of acute rejection within the last 6 months

On stable immunosuppressive therapy for at least 3 months

Ability to provide written informed consent

Willingness and ability to comply with study procedures and sample collection

Exclusion Criteria:

* Use of antibiotics or probiotics within 4 weeks prior to enrollment

Known gastrointestinal disease (e.g. inflammatory bowel disease, celiac disease, short bowel syndrome)

Uncontrolled diabetes mellitus (HbA1c > 9%)

Current infection or active malignancy

Pregnancy or breastfeeding

Participation in another interventional clinical trial within the past 30 days

Known allergy or intolerance to SCFA formulations or study components (lactose intolerance)

Severe hepatic impairment (Child-Pugh class C)

Any condition that, in the opinion of the investigator, may interfere with the participant's ability to complete the study or affect the interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in concentration of serum metabolites after SCFA supplementation | Baseline to Week 12 and Week 12 to washout period
  Quantitative and qualitative changes in the concentration of serum metabolites assessed using targeted metabolomic techniques NMR.
Change in concentration of urine metabolites after SCFA supplementation | Baseline to Week 12 and Week 12 to washout period
  Quantitative and qualitative changes in the concentration of urine metabolites assessed using targeted metabolomic techniques NMR.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) in the contexte of SCFA supplementation | Baseline to Week 12
  Number, type, and severity of AEs assessed through questionnaire, clinical assessment, and lab tests.
Change in inflammatory biomarkers | Baseline to Week 12
  Exploratory analysis of inflammatory markers (CRP, leukocytosis) to assess potential immunomodulatory effects of SCFA.
Changes in estimated glomerular filtration rate (eGFR). | Baseline to Week 12 and Week 24
  Monitoring renal function using eGFR (ml/min/1.73m2) calculated by CKD-EPI.
Tolerability of SCFA supplementation | Baseline to Week 12
  The patient tolerability of SCFA suplementation or placebo assessed through questionnaire.
Change in immunological biomarkers | Baseline to Week 12
  Exploratory analysis of immunological markers (T cell subsets) to assess potential immunomodulatory effects of SCFA.
Changes in urine albumine cretinine ratio (UACR). | Baseline to Week 12 and Week 24
  Monitoring renal function using UACR in the context of using SCFA or placebo.
Changes in the serum level of tacrolimus. | Baseline to Week 12 and Week 24
  Monitoring the serum level of tacrolimus (ng/l) in the context of SCFA supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Martin, Martin, Slovakia, Slovakia